CLINICAL TRIAL: NCT07076641
Title: Phase III, Randomized, Double-blind Study to Assess the Efficacy and Safety of Intravenous Lidocaine Versus Placebo in Patients Receiving Analgesic Morphine Rachi Anesthesia for Major Digestive or Abdominal Surgery by Laparotomy.
Brief Title: Efficacy and Safety of Intravenous Lidocaine Versus Placebo in Patients Receiving Morphine-rachi Analgesia
Acronym: LIDORACHI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-521206-18-00
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Digestive System Disease; Surgery
MeSH Terms: conditions — Digestive System Diseases | interventions — Laparotomy; Morphine

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, comparative, randomized, 2-group parallel, placebo-controlled, double-blind clinical trial
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIDOCAINE Intravenous electric syringe (Experimental): Induction bolus 1.5 mg/kg (adjusted weight) intraoperatively, at the time of anesthetic induction, 15 to 30 min before incision.
  Maintenance 1.5 mg/kg/h until end of care / discharge from the intensive care unit (reduced to 1 mg/kg/h in the post-interventional monitoring room), i.e. between 1 and 2 hours after the end of surgery.
  Interventions: Procedure: rachi morphine anesthesia; Procedure: laparotomy; Drug: Lidocaine IV; Drug: MORPHINE
- PLACEBO Intravenous electric syringe (Placebo Comparator): Induction bolus 1.5 mg/kg (adjusted weight) intraoperatively, at the time of anesthetic induction, 15 to 30 min before incision.
  Maintenance 1.5 mg/kg/h until end of care / discharge from the intensive care unit (reduced to 1 mg/kg/h in the post-interventional monitoring room), i.e. between 1 and 2 hours after the end of surgery.
  Interventions: Procedure: rachi morphine anesthesia; Procedure: laparotomy; Drug: Placebo; Drug: MORPHINE

INTERVENTIONS:
Procedure: rachi morphine anesthesia — Morphine spinal anesthesia is administered before general anesthesia, just after the patient has been admitted to the operating room.
Procedure: laparotomy — major digestive or abdominal surgery by laparotomy
Drug: Lidocaine IV — KABI 20 mg/mL solution for injection (ready-to-use ampoule, no dilution). Each ml of solution contains 20 mg lidocaine hydrochloride (monohydrate form), corresponding to 16.22 mg lidocaine.
  Arms: LIDOCAINE Intravenous electric syringe
Drug: Placebo — Sodium chloride (NaCl) FRESENIUS 0.9% solution for infusion. Each ml contains 9 mg sodium chloride.
  Arms: PLACEBO Intravenous electric syringe
Drug: MORPHINE — The auxiliary drug on which both experimental strategies are based is MORPHINE: Morphine hydrochloride AGUETTANT 0.1 mg/mL Solution for injection (ready-to-use ampoule) for rachi anesthesia.

SUMMARY:
The purpose of this study is to evaluate the superiority of IV lidocaine combined with morphine spinal anesthesia versus placebo combined with morphine spinal anesthesia, in reducing postoperative morphine consumption at 48 hours, in patients undergoing major digestive or abdominal surgery by laparotomy.

DETAILED DESCRIPTION:
This is a prospective, interventional, comparative, randomized, 2-group parallel, placebo-controlled, double-blind, single-center trial designed to evaluate the value of intravenous lidocaine combined with morphine rachi anesthesia in major laparotomy digestive or abdominal surgery.

The study corresponds to a clinical trial of a medicinal product in compliance with Regulation (EU) n°536/2014.

The study population is composed of adult patients receiving morphine spinal anesthesia for major laparotomy surgery and who have signed an informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Major digestive or abdominal surgery (pancreatic, hepatic, colorectal, gynecological, esophageal, gastric, duodenal, small intestine...);
* Scheduled surgery;
* Laparotomy;
* Patient in agreement with morphine rachi anesthesia;
* Social security affiliation;
* Signed informed consent.

Exclusion Criteria:

* Emergency surgery;
* Contraindication to non-steroidal anti-inflammatory drugs: history of gastro duodenal ulcer, renal failure from stage 3 A or higher;
* History of bradycardia and/or known conduction disorder (atrioventricular block) / Pacemaker ;
* Unstable coronary ;
* Myocardial infarction <6 months;
* Severe cardiocirculatory insufficiency;
* Severe hepatic insufficiency;
* Allergy to morphine ;
* Allergy to lidocaine;
* Rhythm disorders at risk of sudden death (e.g. Brugada syndrome);
* Flecaine as usual treatment;
* Chronic pain with level II or III analgesics;
* Gabapentinoids: pregabalin (Lyrica), gabapentin;
* Drug addiction and substitute drugs;
* Epileptic disorders ;
* Myasthenia gravis;
* Creatinine clearance below 10 mL/min;
* Hypokalemia, hypoxia or acid-base disorders;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Inability to understand study information (due to linguistic, psychological, cognitive or literacy problems);
* Women who are or may become pregnant* (of childbearing age, without effective contraception) or who are breast-feeding;
* Patient deprived of liberty, under guardianship or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 2 days
  Total consumption of morphine received postoperatively from the post-interventional monitoring room to 48 hours (in mg) by intravenous and patient-controlled analgesia, and oral dose converted to IV morphine equivalent where applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France